CLINICAL TRIAL: NCT05962138
Title: Characterisation of Pain in Patients With Musculoskeletal Disease: a Prospective, Longitudinal, Observational Study With an Embedded Feasibility Window of Opportunity Sleep Study
Brief Title: A Study of Digital Cognitive Behavioural Therapy for Insomnia in Fibromyalgia
Acronym: Pain-LESS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Big Health Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 252762
Record Dates: First submitted 2023-06-26; First posted 2023-07-27 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2024-08

CONDITIONS: Fibromyalgia
Keywords: sleep; digital; cognitive behavioural therapy for insomnia; fibromyalgia; pain; cognition
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with two parallel study arms: (1) digital cognitive behavioural therapy for insomnia (experimental condition), and (2) treatment as usual (control condition). Randomisation will be using a 1:1 ratio (experimental:control), within minimisation of between group differences in sex, and inclusion status in imaging sub-study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Baseline assessment, randomisation and facilitation of the intervention will be performed by members of the research team who will be blinded to group allocation. The investigators analysing the data will be blinded to group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleepio (dCBT-I) (Experimental): 6-10 weeks of digital cognitive behavioural therapy for insomnia (Sleepio) delivered online.
  Participants will also receive a booklet with general advice for patients with fibromyalgia, including sleep hygiene.
  Interventions: Behavioral: Digital Cognitive Behavioural Therapy for Insomnia
- Treatment as usual (No Intervention): Participants will receive a booklet published by Versus Arthritis designed for patients with fibromyalgia with general advice, including sleep hygiene.

INTERVENTIONS:
Behavioral: Digital Cognitive Behavioural Therapy for Insomnia — 6-10 weeks of digital cognitive behavioural therapy for insomnia (Sleepio) delivered online. In addition participants will receive a booklet published by Versus Arthritis designed for patients with fibromyalgia with general advice, including sleep hygiene.
  Other Names: Sleepio
  Arms: Sleepio (dCBT-I)

SUMMARY:
The goal of this clinical trial is to investigate the potential benefits of a digital Cognitive Behavioural Therapy for Insomnia (dCBT-I) platform, Sleepio, in individuals suffering from fibromyalgia, a condition commonly associated with cognitive issues and sleep disorders.

The main questions this study aims to answer are:

* Does the application of Sleepio improve quality of life in individuals with fibromyalgia?
* Does the use of Sleepio improve cognitive function in individuals with fibromyalgia?
* Does the use of Sleepio enhance sleep quality in these same individuals?
* Does the use of Sleepio improve motor function in this group?

Participants will be randomly assigned to either use the Sleepio platform or standardised health advice, including sleep hygiene material. Those assigned to Sleepio will undergo a series of six 20-minute sessions over 10 weeks with a virtual therapist focusing on cognitive and behavioural strategies for improving sleep.

Participants' quality of life, cognitive function, sleep quality, and pain levels will be monitored and evaluated using online assessment tools. Additionally, a subset of participants will undergo further testing via sleep actigraphy and/or neuroimaging with MRI scans.

Researchers will compare the two groups to determine if the use of Sleepio has a positive effect on quality of life, cognitive function, and sleep quality.

DETAILED DESCRIPTION:
Fibromyalgia patients commonly experience cognitive issues such as concentration and memory difficulties and sleep disorders. Despite the prevalence of these symptoms, no established treatments currently exist. Traditional in-person Cognitive Behavioural Therapy (CBT), which focuses on modifying unhelpful thoughts and behaviours, is both expensive and challenging to deliver on a broad scale. New digital forms of CBT, specifically for insomnia (CBT-I), have shown promise in improving cognitive symptoms and sleep quality, but their effect on fibromyalgia patients is yet to be explored.

The study will investigate the efficacy of 'Sleepio', an established digital CBT-I (dCBT-I) tool. Sleepio has shown effectiveness in treating insomnia and its cognitive symptoms, offering a promising approach to address similar issues in fibromyalgia. Sleepio's approach involves six 20-minute sessions over 10 weeks with a virtual therapist who employs key cognitive and behavioural strategies to enhance sleep quality.

Participants in this study will be randomised in a 1:1 ratio to either treatment with Sleepio treatment or standard care with standard sleep hygiene advice. The primary outcome is quality of life measured on the Revised Fibromyalgia Impact Questionnaire (FIQR), 12 weeks following randomisation. Secondary outcomes include subjective cognition (British Columbia Cognitive Complaints Inventory, BC-CCI), objective cognitive function (tests of reaction time, working memory, processing speed), quantitative cognitive avoidance testing (QCAT), sleep quality (actigraphy, insomnia severity index (ISI), Pittsburgh Sleep Quality Index (PSQI), pain (NRS), fear of movement (Tampa Scale of Kinesiophobia) and quantitative movement assessment. Assessments will be carried out using online tools.

Additionally, a subset of participants will undergo sleep actigraphy and/or neuroimaging using MRI scans for a more detailed analysis.

Primary Objectives:

- Assess the impact of Sleepio (dCBT-I) on quality of life (FIQR) in fibromyalgia patients.

Secondary Objectives:

* Assess the impact of Sleepio (dCBT-I) on subjective (BC-CCI) and objective cognitive function in fibromyalgia patients.
* Investigate the effect of Sleepio on sleep quality (ISI & PSQI) in fibromyalgia patients.
* Investigate cost-effectiveness of Sleepio (dCBT-I)
* Does Sleepio improve subjective and objective measures of motor function in fibromyalgia?

As part of the study, participants will also be invited to join a research database for potential inclusion in future studies conducted by the research group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of fibromyalgia
* Concomitant insomnia, frequent waking in the night or early morning waking
* Self-reported difficulties with concentration or memory
* Reliable internet access

Exclusion Criteria:

* Patients with a poor understanding of English.
* Patients with known neurological or psychiatric conditions (other than depression or anxiety) likely to independently affect the results of pain assessment, for example peripheral diabetic neuropathy in the opinion of the research team
* Major neuropsychiatric disorder (bipolar disorder, schizophrenia or psychotic spectrum disorders)
* Epilepsy
* Cognitive impairment, dementia or neurodegenerative disorder
* Recent or planned surgery
* Current or planned night-time shift work
* Sleep disorders such as sleep apnoea, restless leg syndrome, circadian rhythm disorder, or parasomnia
* Taking prescribed sleep medications on more than 2 nights in past 2 weeks
* Currently receiving other psychological therapy for insomnia
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | 12 weeks
  The revised Fibromyalgia Impact Questionnaire (FIQR), range 0-100, is a self-reported measure designed to assess the overall impact of fibromyalgia on patients' lives, capturing domains such as physical impairment, overall well-being, and the intensity of symptoms like pain, fatigue, stiffness, sleep disturbances, and cognitive problems. Higher scores indicate more severe symptoms.

SECONDARY OUTCOMES:
Change in Revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | 24 weeks
  The revised Fibromyalgia Impact Questionnaire (FIQR), range 0-100, is a self-reported measure designed to assess the overall impact of fibromyalgia on patients' lives, capturing domains such as physical impairment, overall well-being, and the intensity of symptoms like pain, fatigue, stiffness, sleep disturbances, and cognitive problems. Higher scores indicate more severe symptoms.
Sleep quality | 12 weeks
  Changes in sleep pattern on actigraphy between treatment groups
Change in Revised Fibromyalgia Impact Questionnaire (FIQR) from baseline | 52 weeks
  The revised Fibromyalgia Impact Questionnaire (FIQR), range 0-100, is a self-reported measure designed to assess the overall impact of fibromyalgia on patients' lives, capturing domains such as physical impairment, overall well-being, and the intensity of symptoms like pain, fatigue, stiffness, sleep disturbances, and cognitive problems. Higher scores indicate more severe symptoms.
Change in British Columbia Cognitive Complaints Inventory (BC-CCI) from baseline | 12 weeks
  The British Columbia Cognitive Complaints Inventory (BC-CCI), range 0-18, is a rapid screening tool that assesses perceived cognitive difficulties. Higher scores indicate more severe symptoms.
Change in British Columbia Cognitive Complaints Inventory (BC-CCI) from baseline | 24 weeks
  The British Columbia Cognitive Complaints Inventory (BC-CCI), range 0-18, is a rapid screening tool that assesses perceived cognitive difficulties. Higher scores indicate more severe symptoms.
Change in British Columbia Cognitive Complaints Inventory (BC-CCI) from baseline | 52 weeks
  The British Columbia Cognitive Complaints Inventory (BC-CCI), range 0-18, is a rapid screening tool that assesses perceived cognitive difficulties. Higher scores indicate more severe symptoms.
Change in Tampa Scale of Kinesiophobia (TSK) from baseline | 12 weeks
  The Tampa Scale of Kinesiophobia (TSK), range 17-68, is a patient-reported outcome measure designed to quantify kinesiophobia or fear of movement. Higher scores indicate greater fear of movement.
Change in Tampa Scale of Kinesiophobia (TSK) from baseline | 24 weeks
  The Tampa Scale of Kinesiophobia (TSK), range 17-68, is a patient-reported outcome measure designed to quantify kinesiophobia or fear of movement. Higher scores indicate greater fear of movement.
Change in Tampa Scale of Kinesiophobia (TSK) from baseline | 52 weeks
  The Tampa Scale of Kinesiophobia (TSK), range 17-68, is a patient-reported outcome measure designed to quantify kinesiophobia or fear of movement. Higher scores indicate greater fear of movement.
Cost-effectiveness of dCBT-I | 12 weeks
  Health-related quality of life measured with EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version) at baseline, 3- and 6-months. Healthcare resource use data collected at 3- and 6-months. This will be evaluated using cost-effectiveness analysis looking at cost per quality adjusted life year (QALY) with the treatment. QALYs will be estimated using EQ-5D-3L, with higher values indicating better health outcomes. The EQ-5D-3L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease. One quality-adjusted life year (QALY) is equal to 1 year of life in perfect health. QALYs will be calculated by estimating the years of life remaining for a patient following a particular treatment or intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale) from the EQ-5D-3L. Healthcare resource use will be evaluated in the local currency (£).
Cost-effectiveness of dCBT-I | 24 weeks
  Health-related quality of life measured with EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version) at baseline, 3- and 6-months. Healthcare resource use data collected at 3- and 6-months. This will be evaluated using cost-effectiveness analysis looking at cost per quality adjusted life year (QALY) with the treatment. QALYs will be estimated using EQ-5D-3L, with higher values indicating better health outcomes. The EQ-5D-3L is a generic tool for Patient Reported Outcomes (PRO) measurement that can assess patients' quality of life, irrespective of the disease. One quality-adjusted life year (QALY) is equal to 1 year of life in perfect health. QALYs will be calculated by estimating the years of life remaining for a patient following a particular treatment or intervention and weighting each year with a quality-of-life score (on a 0 to 1 scale) from the EQ-5D-3L. Healthcare resource use will be evaluated in the local currency (£).
Changes in brain structure | 12 weeks
  Change in brain grey matter volume on structural MRI
Changes in brain functional connectivity | 12 weeks
  Changes in brain resting state functional connectivity on resting-state functional MRI
Changes in neurotransmitter concentration in the insular | 12 weeks
  Changes in neurotransmitter concentration in the insular on magnetic resonance spectroscopy
Changes in brain function | 12 weeks
  Changes in brain resting state activity on arterial spin labelling (ASL) on brain MRI

CONTACTS AND LOCATIONS:
Overall Officials: Anushka Soni, Dr, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified data are available upon reasonable request
Supporting Information: Study Protocol
Time Frame: Following publication of results
Access Criteria: Available upon reasonable request

DOCUMENTS (3):
  • Study Protocol (2023-02-07): https://cdn.clinicaltrials.gov/large-docs/38/NCT05962138/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/38/NCT05962138/SAP_001.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT05962138/ICF_002.pdf